CLINICAL TRIAL: NCT06162949
Title: Vonoprazan-based Triple Therapy vs. Standard Triple Therapy for Helicobacter Pylori Eradication in Adolescents: A Randomized, Double-blinded Controlled Trial
Brief Title: Vonoprazan for Helicobacter Pylori Eradication in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sameh A. Lashen, Assistant Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0306381
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Treatment Effectiveness
Keywords: Helicobacter pylori; Vonoprazan; Standard triple therapy; Adolescent; Eradication rate
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonoprazan-based triple therapy (Experimental): Vonoprazan tablets 20 mg twice daily plus Amoxicillin 50 mg/kg/day capsules or suspension [maximum daily dose 2 g] plus Clarithromycin 20 mg/kg/day tablets or suspension [maximum daily dose 1 g] The triple combination will be given for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Clarithromycin
- Proton pump-based triple therapy "standard triple therapy" (Active Comparator): Esomeprazole tablets [20 mg/day if < 30 kg and 40 mg/daily if ≥ 30 kg] on two divided daily doses plus Amoxicillin 50 mg/kg/day capsules or suspension [maximum daily dose 2 g] plus Clarithromycin 20 mg/kg/day tablets or suspension [maximum daily dose 1 g] The triple combination will be given for 14 days
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan — an acid suppressor therapy that inhibits the H+, K+-ATPase enzyme system in a potassium-competitive manner.
  Other Names: Vonacidan; Tavoniza; Vondalous
  Arms: Vonoprazan-based triple therapy
Drug: Amoxicillin — An antibiotic of penicillins antibiotic group
  Other Names: Emox; Ibiamox; Amoxicid
Drug: Clarithromycin — An antibiotic of macrolide group
  Other Names: Klacid; Klarithro; Klarimix; Infectocure
Drug: Esomeprazole — An acid suppressor therapy that blocks the proton pump.
  Other Names: Nexium; Neximash; Esomium; Nexicure
  Arms: Proton pump-based triple therapy "standard triple therapy"

SUMMARY:
The trial tends to evaluate the efficacy of vonoprazan-based triple therapy in eradicating H. Pylori infection in adolescent patients in Egypt, in comparison to standard treatment regimens to determine if it offers superior eradication rates (VONTAPE trial).

DETAILED DESCRIPTION:
The VONTAPE trial will compare two treatment regimens for Helicobacter pylori eradication among adolescent patients presented to the gastroenterology department in an Egyptian institute. the eligible subjects will be randomly assigned to one of the two protocols (vonoprazan based vs. proton pump inhibitor-based triple therapy) for two weeks. then the eradication rates will be compared between the two study groups to see if there is a difference in efficacy.

The currently available eradication regimens in our country show a low to intermediate eradication rate (50-75%). At the same time, H. pylori infection is prevalent.

Recently, the FDA approved vonoprazan-based regimens for adult H. pylori infection with high eradication rates even in the settings of clarithromycin antibiotic resistance.

In the VOTSAPE trial, we will test this efficacy in the < 18 years adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Children in the age group (10-18 years), both genders, referred with dyspeptic complaints such as heartburn, dyspepsia, nausea, and epigastric pain.
2. Who is positive for H. Pylori infection by a standardized diagnostic test.
3. Pediatric patients with a clinical, laboratory, and endoscopic diagnosis of H.P.-positive gastritis and the other conditions necessary for H.P. eradication according to the Maastricht V consensus report.

Exclusion Criteria:

1. allergy to any of the drugs used in the study
2. previous attempts to eradicate H.P.
3. Use of antibiotics, acid-suppression, bismuth, or probiotics 4 weeks before enrollment.
4. Children with conditions that affect medication absorption e.g. celiac or Crohn's disease.
5. Liver or kidney failure.
6. symptoms suggestive of functional disorders.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 242 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Helicobacter Pylori eradication rate | 4 weeks after completion of treatment
  Number of patients who will test negative for H. pylori after treatment completion.

SECONDARY OUTCOMES:
The adverse events during therapy | During the treatment duration, and the end of the 2 weeks treatment protocol
  Treatment-related adverse effects (TRAEs) such as abdominal discomfort, diarrhea, vomiting, nausea, flatulence, taste disturbance, or loss of appetite, the need for discontinuation of the H. pylori therapy; and/or headache.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh A Lashen, MD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lashen SA, Shamseyea MM, Metwally RH, Abou-Farrag G, Elkaragy ES. Vonoprazan-Based Triple Therapy Versus Esomeprazole-Based Triple Therapy for H. pylori Eradication in Adolescents (VONTAPE): A Randomized, Double-Blind Controlled Trial. Helicobacter. 2025 Sep-Oct;30(5):e70083. doi: 10.1111/hel.70083. PMID 41131746